CLINICAL TRIAL: NCT05559632
Title: Peri-Implant Marginal Bone Loss And Implant Stability In Maxillary Implant Overdenture When Using Osseodensification Versus Conventional Drills: A Randomized Clinical Trial
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Collaborators: prof. Nadia Ahmed Abbas (Unknown); dr. Doaa Mahmoud abd elhameed elkady (Unknown)
Responsible Party: Principal Investigator, Marwa Essam El-Dein Mohamed, lecture assistant, Cairo University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 13722
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Completely Edentulous Maxilla; Implant Placement; Maxillary Implant Overdenture
MeSH Terms: interventions — Osteotomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional drilling group (Active Comparator): drilling the other contralateral sites of bone using the conventional sequential drilling system according to the manufactural instruction.
  Interventions: Procedure: osteotomy for implant placement
- osseodensification drilling group (Experimental): bone preparation was performed using tapered multifluted burs (Densah Bur; Versah, MI, USA) at 800- 1200 rpm counterclockwise rotation under saline irrigation. Drilling to the desired depth using the tapered densah pilot drill with speed of 800-1200 rpm with copious irrigation without any lateral pressure with clock wise motion.
  Interventions: Procedure: osteotomy for implant placement

INTERVENTIONS:
Procedure: osteotomy for implant placement — preparing the bone for implant placement

SUMMARY:
Is to compare between the conventional drills versus osseodensification drills for implant stability and peri-implant marginal bone loss in maxillary implant overdenture.

DETAILED DESCRIPTION:
Comprehensive clinical examination and understanding of patient's chief complaints and their expectations from the prosthesis.

* medical and dental history
* A complete denture will be constructed for each patient to aid in the scan technique, if the patient has an denture, it will be evaluated to be used.
* The complete denture will be constructed following conventional denture fabrication procedures.
* CBCT radiograph will be taken for bone height and width, and identify the vital structures before implant placement.
* A surgical guide will be used to aid in the implant placement, each patient will be scheduled for surgery to insert four root form implants. Each patient will receive four implants at canine and premolar regions from the same implant manufacturer.

Study group: The osseodensification drilling group (G1), bone preparation was performed using tapered multifluted burs (Densah Bur; Versah, MI, USA) at 800- 1200 rpm counterclockwise rotation under saline irrigation. Drilling to the desired depth using the tapered densah pilot drill with speed of 800-1200 rpm with copious irrigation without any lateral pressure with clock wise motion.

Control group: In the conventional drilling group (G2), drilling the other contralateral sites of bone using the conventional sequential drilling system according to the manufactural instruction.

* All patients received 2gm/day amoxicillin, clavulanate and 50 mg/8 hours non-steroidal anti-inflammatory analgesics for 5 days postoperatively. Postoperative instructions included a soft diet and appropriate oral hygiene measures with 0.2% chlorhexidine mouth rinse.
* After four months, the implants will be exposed and attachment (stud attachment) will be screwed to the implants. Then, overdenture pick-up is done. * Number of visits & follow up period

  * 5 visits for construction of denture
  * 1 visit for CBCT
  * 1 visit for implant insertion
  * 1 visit for attachment placement and pick-up of overdenture
  * Patients will be recalled at base line,4 and 7 weeks 4 and 12 months following implant insertion for outcomes assessment

ELIGIBILITY:
Inclusion Criteria:

1. Patients with completely edentulous maxilla.
2. Sufficient inter-arch space not less 13mm inter-arch space.
3. sufficient bone height to allow usage of at least 10mm implant length.
4. Normal maxilla-mandibular relationship.
5. minimum radiographic bone width bucco-palatally in canine and premolar regions to place at least 3.5mm implant diameter.
6. participants more than forty years old.
7. Opposing fully or partially restored dentition.

Exclusion Criteria:

* 1- Skeletal mal-relation. 2- Unmotivated patients to maintain adequate oral hygiene to follow up. 3- Patients with neuromuscular and Psychiatric disorders. 4- Systematic disease affecting bone and periodontal health such as diabetic patients.

  5- Insufficient inter-arch space less than 13mm. 6- Patients with physical reasons that could affect follow up. 7- patients administrating antibiotics 8- smoker patients 9- patients with any systemic or local condition that obstacles implant placement 10- patients with a history of radiotherapy in the head and neck region

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Peri-implant marginal bone loss | 1 year
  Radiographic follow up will be performed for marginal bone loss. Serial of standardized digital periapical radiographs using; long cone paralleling technique, XCP periapical film holder and an individually constructed radiographic acrylic template will be taken at the time of implant placement (base line) then at 4,12 months.

SECONDARY OUTCOMES:
Implant stability measurements | 4 months
  The Osstell will be used according to the manufacturer's instructions and held perpendicular to the provided implant smart peg. Osstell values (ISQ) are going to be obtained for the bucco-lingual, mesio-distal surfaces of each implant. Three measurements will be made for each surface and the mean will be obtained for statistical analysis.for each implant will be done at the time of surgery, at 4 weeks , 7weeks and 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry- Cairo university, Cairo, Egypt